CLINICAL TRIAL: NCT05668676
Title: Effect of Short-Term Prednisone Therapy on C-Reactive Protein Change in Emergency Department Patients With Acute Heart Failure and Elevated Inflammatory Marker
Brief Title: Effect of Short-Term Prednisone Therapy on C-Reactive Protein Change in Emergency Department Patients With Acute Heart Failure and Elevated Inflammatory Markers ( CORTAHF )
Acronym: CORTAHF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220428; 2022-001604-17 (EudraCT Number)
Record Dates: First submitted 2022-11-21; First posted 2022-12-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; Emergency Department; Prednisone therapy
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental)
  Interventions: Drug: Prednisone arm
- Control group (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Prednisone arm — 2 tabs of 20 mg prednisone per day during 7 days added to usual care medications
  Arms: Interventional group
Other: Usual care — Usual care alone as per European guidelines, which includes oxygen in case of hypoxia, low dose furosemide (40mg or daily dosage), and iv nitrates if no contra-indication.
  Arms: Control group

SUMMARY:
Acute heart failure (AHF) is a common discharge diagnosis in the emergency department (ED), associated with 1-month mortality of 6%, and a 30% risk rate of 1-month rehospitalisation. Current guidelines recommend the use of nitrates and low dose diuretics to treat congestion, but to date, no drug has ever shown any improved clinical outcome when given at the acute phase.

Several studies suggest that there is a high inflammatory component in AHF, with elevated markers such as IL6 and C-reactive protein (CRP). As it is the case in other acute respiratory disease, a short course of steroid therapy may limit the inflammatory response and in turn, improve AHF prognosis.

The objective of the study is to assess the effect of a 7-day course of steroid introduced in the ED on inflammatory response

DETAILED DESCRIPTION:
A multicentric (5 EDs in France), phase 3, comparative, open-label, randomised controlled study in 2 parallel-group comparing usual AHF treatment (control group) with usual AHF treatment + prednisone (intervention group). The objective is to assess the effect of a 7-day course of prednisone therapy started in the ED and continued for up to 7 days on the change of CRP level.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years of age
2. Unplanned ED visit within the 12 hours prior to Screening with acute or worsening dyspnea and/or orthopnea, and Pulmonary congestion on chest X-ray or lung ultrasound.
3. All measures from presentation to randomization of systolic blood pressure ≥ 100 mmHg, and of heart rate ≥ 60 bpm.
4. Written informed consent to participate in the study.
5. Affiliation to a french social security system (beneficiary or legal)
6. Biomarker levels indicative of congestion and inflammation: At Screening, NT-proBNP > 1,500 pg/mL or BNP>375 pg/mL and CRP > 40 mg/L
7. Patient agrees for follow-up visit at the hospital at day 7 in case of earlier discharge and Day 30.

Exclusion Criteria:

1. Anticipated life expectancy less than 6 months
2. Mechanical ventilation (not including CPAP/BIPAP) prior to Screening.
3. Significant pulmonary disease contributing substantially to the patients' dyspnea such as FEV1< 1 liter or need for chronic systemic or non- systemic steroid therapy, or any kind of primary right heart failure such as primary pulmonary hypertension or recurrent pulmonary embolism.
4. Myocardial infarction, unstable angina or cardiac surgery within 3 months, or cardiac resynchronization therapy (CRT) device implantation within 3 months, or percutaneous transluminal coronary intervention (PTCI), within 1 month prior to inclusion.
5. Index Event (admission for AHF) triggered primarily by a correctable etiology such as significant arrhythmia (e.g., sustained ventricular tachycardia, or atrial fibrillation/flutter with sustained ventricular response >130 beats per minute, or bradycardia with sustained ventricular arrhythmia <45 beats per minute), infection, severe anemia, acute coronary syndrome, pulmonary embolism, exacerbation of COPD, planned admission for device implantation or severe non-adherence leading to very significant fluid accumulation prior to admission and brisk diuresis after admission. Troponin elevations without other evidence of an acute coronary syndrome are not an exclusion.
6. Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
7. History of heart transplant or on a transplant list, or using or planned to be implanted with a ventricular assist device.
8. Sustained ventricular arrhythmia with syncopal episodes within the 3 months prior to screening that is untreated.
9. Presence at screening of any hemodynamically significant valvular stenosis or regurgitation, except mitral or tricuspid regurgitation secondary to left ventricular dilatation, or the presence of any hemodynamically significant obstructive lesion of the left ventricular outflow tract.
10. Primary liver disease considered to be life threatening (defined by a prothrombin time < 30%)
11. eGFR < 30 mL/min/1.73m2 or eGFR > 80 mL/min/1.73m2 (as estimated by the simplified MDRD formula) at inclusion or history of dialysis.
12. Systemic steroid therapy, within 30 days from inclusion.
13. Inability to consent, or patient under guardianship measure
14. Participation in another intervention trial in the past 30 days
15. Anticipated non-adherence to study protocol or follow-up.
16. Pregnant or nursing (lactating) women.
17. Known hypersensitivity to steroids or constituents of prednisone tablets (excipients)
18. Psychotic states not yet controlled by treatment
19. Concomitant administration of live vaccines and up to 3 months before end of corticotherapy administration
20. Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom
21. Persons subject to psychiatric care without their consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change in CRP value from inclusion to day 7 | Day 7
  To assess the effects of prednisone therapy started in the ED and continued for up to 7 days on the change of CRP level.

SECONDARY OUTCOMES:
The composite of death, or hospital readmission for decompensated HF through day 30 or worsening heart failure occurring between 24h after randomization through the earliest of discharge or day 7 | Day 30
Comparisons on the effects on change in quality of life | Day 7
  Changes in quality of life measured by the EQ-5D-5L from randomization to day 7
Comparisons on the effects on change in quality of life | Day 30
  Changes in quality of life measured by the EQ-5D-5L from randomization to Day 30
Symptoms of heart failure | Day 7
  Changes in symptoms of congestion (NYHA classification, orthopnea, peripheral edema, rales, jugular venous pulse, dyspnea) at day 7
signs of heart failure | Day 7
  Changes in heart failure signs
Change in weight from randomization to day 7 | Day 7
Death from any cause at day 30 | Day 30
Readmission for HF or death | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan FREUND, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided